CLINICAL TRIAL: NCT06452069
Title: A Multicentre, Randomised, Prospective Study Investigating the Efficacy and Safety of an Essential Oil-Based Preparation Administered to Mild and Moderately Severe COVID-19 Positive Patients
Brief Title: Efficacy and Safety Study of Essential Oil-Based Preparation Administered to COVID-19 Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biodex S.A (Industry)
Collaborators: Gama CRO Tıbbi IIac Arastirma Org.Tic.Ltd.Sti (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC2021-ID19
Record Dates: First submitted 2024-06-06; First posted 2024-06-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: COVID-19 Respiratory Infection; COVID-19
Keywords: Essential Oil, antiviral, Main Protease, COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Prospective Study
Who Masked: Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1: (n=140) Investigational Product 10 ml, drinkable ampoule (1 ampoule) (1 time only)
  Interventions: Other: IMMUNO19
- Group 2 (Placebo Comparator): Group 2: (n=140) Placebo 10 ml (1 ampoule) (1 time only)
  Interventions: Other: IMMUNO19

INTERVENTIONS:
Other: IMMUNO19 — 280 participants will be divided into 2 groups. There will be 140 participants in the groups.
  The 1st group will receive IMMUNO19 10 mL one time, The 2nd group will receive Placebo 10 mL for one time.
  Other Names: Essential Oils Combination

SUMMARY:
The aim of this study was to compare the efficacy and safety of the essential oil-based product in patients with mild to moderate symptomatic COVID-19 Positive infection confirmed by PCR. A computational simulation approach of the molecular interaction (binding) of the main components of essential oils exhibiting antiviral activity with known intracellular protein targets of SARS-CoV-2 (nsp5: Main Protease) was adopted as a rationale for this study. SARS-CoV-2, a single-stranded RNA virus, has four major structural proteins Spike (S), Membrane (M), Envelope glycoprotein (E) and Nucleocapsid (N) protein and non-structural proteins (nsp). These non-structural proteins, of which there are 16 in total in the genome of the virus, play key roles in the mechanisms of the virus life cycle, including replication, transcription, protein synthesis and modification of RNA. Main protease (Main protease, Mpro, 3CLpro), virus Since they are directly involved in the maturation of these nsp proteins, which have an important role in many mechanisms of the life cycle, they have been the target enzyme in the development of new antiviral drugs for the treatment of COVID-19. In this study, our main rationale is to investigate the effect of essential oils on nsp5: Main Protease enzyme activations.

DETAILED DESCRIPTION:
The indiscriminate use of antimicrobial agents has led to the emergence of a number of drug-resistant bacteria, fungi and viruses. To overcome the increasing resistance of pathogenic microbes, more effective antimicrobial agents with new modes of action must be developed.

Medicinal plants used in traditional medicines to treat infectious diseases are an abundant source of new bioactive secondary metabolites. Therefore, in the last few years, various medicinal plants and plant extracts have been screened for their antimicrobial activities . Essential oils obtained from aromatic medicinal plants (e.g. fennel (Foeniculum vulgare), mint (Mentha piperita), thyme (Thymus vulgaris)) have been shown to have antimicrobial activity against gram-positive and gram-negative bacteria as well as yeasts, It has been reported to be active against fungi and viruses. They are mixtures of different lipophilic and volatile substances such as monoterpenes, sesquiterpenes and/or phenylpropanoids and have a pleasant odour. They are also part of the pre-formed defence system of higher plants are thought to be . Monoterpenes have been widely studied, especially for their antiviral properties.

Nowadays, the use of essential oils is becoming increasingly widespread both in pharmacies and in various stores. The use of essential oils for therapeutic purposes is expanding. The molecules that make up certain essential oils have shown various antiviral properties:

* Either by neutralising the virus before it enters the cell,
* By changing the capsid or envelope of the virus,
* Either by binding to receptors used by viruses and preventing their access to cells.

Herbal products are an important source of herbal remedies and other medicines. Essential oils have shown various pharmacological activities, such as antiviral activity, and have therefore been implicated in SARS-CoV- It has been suggested to have potential activity against 2. Essential oils can easily penetrate the viral membrane due to their lipophilicity and can cause rupture of the viral membrane.

In addition, crude essential oils often have many active components that can act on different parts of the virus, including cell entry, translation, transcription and assembly. Anti-inflammatory, immune regulation on the respiratory system of the host, have other beneficial pharmacological effects, including bronchiectasis and mucolytics.

Essential oils have many advantages because they promise volatile antiviral molecules, making them useful either alone or in combination with other chemotherapeutic drugs, making them potential drug targets for the prevention and treatment of COVID-19.

In this study, a computational simulation approach of the molecular interaction (binding) of the main components of essential oils exhibiting antiviral activity with known intracellular protein targets of SARS-CoV-2 (nsp5: Master Protease) was adopted as a rationale. A single-chain.

The RNA virus SARS-CoV-2 has four main structural proteins Spike (S), Membrane (M), Envelope glycoprotein (E) and Nucleoapsid (N) proteins and non-structural proteins (nsp) .

These non-structural proteins, of which there are 16 in total in the genome of the virus, play a key role in the mechanisms of the virus life cycle, including replication, transcription, protein synthesis and modification of RNA. Main protease (Mpro, 3CLpro) has been the target enzyme for the development of new antiviral drugs for the treatment of COVID-19 , as they are directly involved in the maturation of these nsp proteins, which have an important role in many mechanisms of the virus life cycle. Our main rationale in this study is to investigate the effect of essential oils on nsp5: Main Protease enzyme activations.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 18<X< 65 years of age.
* The participant must be willing and able to give written informed consent. The volunteer must provide his/her consent on his or her behalf, a legally acceptable representative (i.e., an International Harmonization Council [ICH] and adopted by local law as appropriate can be used) must give informed consent on his/her behalf.
* PCR test COVID-19 positive diagnosis and mild to moderate disease stage is required.
* The participant must agree not to receive vaccines administered for COVID-19 during the study.

Exclusion Criteria:

* Patients < 18 years of age,
* Positive diagnosis of severe COVID-19 with symptoms of basic severity: patients with respiratory distress, signs of mental confusion and impaired consciousness that develop depending on the severity of the stage of the disease,
* Patients on active antiviral therapy,
* Patients with creatine clearance < 30 ml/min and renal impairment,
* NYHA III-IV, Stage D heart failure patients requiring frequent hospitalization,
* Uncontrolled coagulopathy,
* Patients with advanced liver failure,
* Patients with active infections such as hepatitis B, hepatitis C and HIV, diseases requiring systemic treatment,
* Patients with active malignancy and known history of cancer,
* Those who do not have sufficient psychic state to disrupt working rounds,
* Active drug users,
* Known hypersensitivity and allergic reaction to the components of the preparation,
* Current participation in another interventional treatment study with an investigational agent,
* Recent use of the investigational product within 28 days of the first dose of the investigational product use or presence of a research device during screening,
* Pregnant or breastfeeding women,
* Patients who did not give written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Clinical and virological cure rate in patients with PCR-confirmed mild to moderate symptomatic COVID-19 Positive infection treated with an essential oil-based product | 0th Day
  Day 0 Participant symptoms and quantitative PCR of viral load
Clinical and virological cure rate in patients with PCR-confirmed mild to moderate symptomatic COVID-19 Positive infection treated with an essential oil-based product | 2nd Day
  Day 2 Participant symptoms
Clinical and virological cure rate in patients with PCR-confirmed mild to moderate symptomatic COVID-19 Positive infection treated with an essential oil-based product | 6th Day
  Day 6 Participant symptoms and quantitative PCR of viral load
Clinical and virological cure rate in patients with PCR-confirmed mild to moderate symptomatic COVID-19 Positive infection treated with an essential oil-based product | 10th Day
  Day 10 Participant symptoms and quantitative PCR of viral load
TClinical and virological cure rate in patients with PCR-confirmed mild to moderate symptomatic COVID-19 Positive infection treated with an essential oil-based product. | 20th Day
  Day 20 Participant symptoms and quantitative PCR of viral load
Clinical recovery defined by the absence of clinical signs of infection | 0th Day
  Clinical signs of acute respiratory infection disappearance (cough and difficulty breathing),Fever within normal temperature ranges, clinical improvement, although the participant has pseudo-symptoms
Clinical recovery defined by the absence of clinical signs of infection | 2nd Day
  Clinical signs of acute respiratory infection disappearance (cough and difficulty breathing),Fever within normal temperature ranges, clinical improvement, although the participant has pseudo-symptoms
Clinical recovery defined by the absence of clinical signs of infection | 6th Day
  Clinical signs of acute respiratory infection disappearance (cough and difficulty breathing),Fever within normal temperature ranges, clinical improvement, although the participant has pseudo-symptoms
Clinical recovery defined by the absence of clinical signs of infection | 10th Day
  Clinical signs of acute respiratory infection disappearance (cough and difficulty breathing),Fever within normal temperature ranges, clinical improvement, although the participant has pseudo-symptoms
Clinical recovery defined by the absence of clinical signs of infection | 20th Day
  Clinical signs of acute respiratory infection disappearance (cough and difficulty breathing),Fever within normal temperature ranges, clinical improvement, although the participant has pseudo-symptoms
Aggravation of the clinical picture | 0th Day
  Appearance of a new sign that was not present at the beginning (not requiring hospitalization),Indicator of hospitalization during the study period,Hospitalization,Hospitalization with oxygen requirement,Hospitalization in intensive care, Death due to COVID-19
Aggravation of the clinical picture | 2nd Day
  Appearance of a new sign that was not present at the beginning (not requiring hospitalization),Indicator of hospitalization during the study period,Hospitalization,Hospitalization with oxygen requirement,Hospitalization in intensive care, Death due to COVID-19
Aggravation of the clinical picture | 6th Day
  Appearance of a new sign that was not present at the beginning (not requiring hospitalization),Indicator of hospitalization during the study period,Hospitalization,Hospitalization with oxygen requirement,Hospitalization in intensive care, Death due to COVID-19
Aggravation of the clinical picture | 10th Day
  Appearance of a new sign that was not present at the beginning (not requiring hospitalization),Indicator of hospitalization during the study period,Hospitalization,Hospitalization with oxygen requirement,Hospitalization in intensive care, Death due to COVID-19
Aggravation of the clinical picture | 20th Day
  Appearance of a new sign that was not present at the beginning (not requiring hospitalization),Indicator of hospitalization during the study period,Hospitalization,Hospitalization with oxygen requirement,Hospitalization in intensive care, Death due to COVID-19
Virological evaluation | 0th Day
  Qualitative PCR Test and Quantitative PCR Test
Virological evaluation | 6th Day
  Qualitative PCR Test and Quantitative PCR Test
Virological evaluation | 10th Day
  Qualitative PCR Test and Quantitative PCR Test
Virological evaluation | 20th Day
  Qualitative PCR Test and Quantitative PCR Test

SECONDARY OUTCOMES:
Evaluation of time from inclusion to recovery in days | 0th Day
  Negative PCR and viral load
Evaluation of time from inclusion to recovery in days | 6th Day
  Negative PCR and viral load
Evaluation of time from inclusion to recovery in days | 10th Day
  Negative PCR and viral load
Evaluation of time from inclusion to recovery in days | 20th Day
  Negative PCR and viral load
Incidence of adverse events and serious advers event | 0th Day
  Collection of adverse events and serious adverse events
Incidence of adverse events and serious advers event | 2nd Day
  Collection of adverse events and serious adverse events
Incidence of adverse events and serious advers event | 6th Day
  Collection of adverse events and serious adverse events
Incidence of adverse events and serious advers event | 10th Day
  Collection of adverse events and serious adverse events
Incidence of adverse events and serious advers event | 20th Day
  Collection of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kanat Tayfun, MD, Principal Investigator — Bagcilar Training and Research Hospital
Locations (10):
- Turkey (Türkiye) (10):
  - Bağcılar Training and Research Hospital, Istanbul, Bagcılar
  - Gaziosmanpaşa Training and Research Hospital, Istanbul, Gaziosmanpaşa
  - Kocaeli City Hospital, Kocaeli, İzmit
  - Göztepe Süleyman Yalçın City Hospital, Istanbul, Kadıköy
  - Kartal Dr. Lütfi Kırdar City Hospital, Istanbul, Kartal
  - Akdeniz University, Antalya, Konyaaltı
  - Süreyyapaşa Chest Disease and Thoracic Surgery Training and Research Hospital, Istanbul, Maltepe
  - Umraniye Training and Research Hospital, Istanbul, Umraniye
  - Antalya Atatürk Public Hospital, Antalya
  - Cemil Taşcıoğlu City Hospital, Istanbul, Şişli